CLINICAL TRIAL: NCT05073016
Title: The Effect of Intermittent Theta Burst Stimulation on Motor Learning in Healthy Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Medeniyet University (Other)
Collaborators: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Esma Nur KOLBAŞI, Researcher, Istanbul Medeniyet University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: IstanbulMU21
Record Dates: First submitted 2021-10-07; First posted 2021-10-11 (Actual); Last update posted 2022-03-02 (Actual); Status verified 2022-02

CONDITIONS: Healthy
MeSH Terms: interventions — Transcutaneous Electric Nerve Stimulation

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Finger Taping Task + iTBS intermittent group (Active Comparator): Finger Taping Task + iTBS Daily application group: the group receives these applications every other day for 5 sessions.
  Interventions: Other: neuromodulation
- Finger Taping Task intermittent Group (Active Comparator): Finger Taping Task intermittent application group: the group receives the application every other day for 5 sessions.
  Interventions: Other: motor learning training

INTERVENTIONS:
Other: neuromodulation — neuromodulation: Neuromodulation is technology that acts directly upon nerves. It is the alteration-or modulation-of nerve activity by delivering electrical or magnetic stimulus/current.
  Arms: Finger Taping Task + iTBS intermittent group
Other: motor learning training — motor learning training requires performing a sequential training called finger taping task
  Arms: Finger Taping Task intermittent Group

SUMMARY:
This study investigates the effect of different application frequencies of intermittent theta burst stimulation on motor learning in healthy adults.

ELIGIBILITY:
Inclusion Criteria:

* being at the age of 40-75 years

Exclusion Criteria:

* visual disability
* cognitive or psychiatric problems such as dementia, depression, etc.

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2021-11-01 (Actual); Primary Completion 2022-02-04 (Actual); Study Completion 2022-02-05 (Actual)

PRIMARY OUTCOMES:
Finger Taping Task | 5 minutes
  The total right answers and the mean response time in the finger taping task will be recorded

CONTACTS AND LOCATIONS:
Overall Officials: Burcu Ersöz Hüseyinsinoğlu, PhD, Study Director — Istanbul University - Cerrahpasa
Locations (1):
- İstanbul Bakırköy Ruh ve Sinir Hastalıkları Hastanesi, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No